CLINICAL TRIAL: NCT06869733
Title: Effects of Scooping Mobilization With and Without Scapulothoracic Mobilization in Pain Range of Motion and Activities of Daily Living in Patients of Lateral Epicondylalgia
Brief Title: Scooping Mobilization With and Without Scapulothoracic Mobilization in Patients of Lateral Epicondylalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/24/0125
Record Dates: First submitted 2025-03-04; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Lateral Epicondylitis
Keywords: Scooping mobilization; scapulothoracic mobilization; activities of daily livings; lateral epicondylalgia
MeSH Terms: conditions — Tennis Elbow

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Scooping Mobilization (Active Comparator): Group A treated with scooping mobilization only.
  Interventions: Other: Scooping Mobilization
- Scooping Mobilization with Scapulothoracic mobilization (Experimental): Group B treated with scooping mobilization with scapulothoracic mobilization.
  Interventions: Other: Scooping Mobilization with Scapulothoracic mobilization

INTERVENTIONS:
Other: Scooping Mobilization — Group A treated with only scooping mobilization with frequency of 2 to 3 times in a week for consecutive 4 weeks.
  Arms: Scooping Mobilization
Other: Scooping Mobilization with Scapulothoracic mobilization — Group B treated with scooping mobilization with scapulothoracic mobilization, which was given 2 to 3 times in a week for consecutive 4 weeks.
  Arms: Scooping Mobilization with Scapulothoracic mobilization

SUMMARY:
Lateral epicondylalgia is well known musculoskeletal disorder now a day. Lateral epicondylalgia is a disorder in which pain and tenderness at lateral part of elbow. This study is targeting the scapulothoracic mobilization and scooping mobilization at lateral epicondylalgia. This study is single-blinded Randomized Clinical Trial will be conducted in Fatima memorial Hospital and Bajwa hospital Lahore. Non-probability convenience sampling will be used with 38 Participants involved in this study is with age of 18 to 45 with presence of pain and tenderness around lateral epicondyle, positive Cozens test and maudsley test, scapular dyskinesia, pain on resisted elbow extension, wrist extension and gripping activities. In this study, one group is treated with scooping mobilization with scapulothoracic mobilization. Second group is treated with scooping mobilization alone. The participants will be randomized into two Groups by computer generated randomization software. Outcomes measures which are used in this study is Numeric pain rating scale for pain, goniometer for range of motion and patient related tennis elbow evaluation for activities of daily livings for patients of lateral epicondylalgia.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-40 years
* Pain and tenderness around lateral epicondyle
* Pain on resisted elbow extension ,wrist extension and gripping activities
* Gender both male and female.
* Scapular Dyskinesia.
* Positive Cozen test and maudsley test for lateral epicondylalgia.
* With moderate pain intensity on Numeric Pain Rating Scale (NPRS) with a score of 3 or higher

Exclusion Criteria:

* Any injury or disease around the shoulder, elbow and wrist on affected side
* Cervical radiculopathy.
* Local steroid injection
* History of fracture of humerus, radius, ulna which is affected upper extremity

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 38 (Actual)
Dates: Start 2023-05-02 (Actual); Primary Completion 2023-12-23 (Actual); Study Completion 2024-07-02 (Actual)

PRIMARY OUTCOMES:
Patient Related Tennis Elbow Evaluation Scale | 4th weeks
  It consist of two subscales, one is pain and second is functional subscale (specific activities: 6 and usual activities . The pain scale is scored out of 50 by summing five items. The function subscale (six items) and usual function subscale (four items) are summed divided by two to create the Function Subscale. The pain score is added to the function score to determine the final score. A score of 100 indicates the highest level of commitment, while a score of 0 indicates no involvement at all..
Numeric Pain Rating Scale | 4th weeks
  It rates from 0 to 10. 0 means no pain while 10 means maximum pain.
Range of Motion of Elbow | 4th weeks
  Goniometer is to check ranges of elbow flexion and extension
Range of Motion of Wrist | 4th weeks
  Goniometer is to check ranges of wrist flexion and extension
Readings of scapulometer to measure scapular dyskinesia in cm | 4th weeks
  The medial boundary and inferior angle prominence in relation to the thorax can be measured with a Scapulometer. The minimal detectable change (MDC) was determined to be 1.2-1.3 mm.

CONTACTS AND LOCATIONS:
Overall Officials: Humera Mubashar, MSOMPT, Principal Investigator — Riphah International University
Locations (2):
- Pakistan (2):
  - Dr. Humera Mubashar, Lahore, Punjab Province
  - Dr. Faiza Amjad, Lahore, Punjab Province

IPD SHARING:
Plan to Share IPD: No